CLINICAL TRIAL: NCT02447107
Title: The Utilization of Mobile Phone Technology to Quantitatively Assess Functional Outcomes of Chronic Pain Patients- A Feasibility Study
Brief Title: Mobile Phone Technology for Chronic Pain Patients- A Feasibility Study
Status: Terminated | Type: Observational
Why Stopped: Study feasibility issues
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1409015460
Record Dates: First submitted 2015-05-13; First posted 2015-05-18 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Technology; Mobile Phone Applications
MeSH Terms: conditions — Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Outpatients: Outpatients enrolled in this study are required to complete study assessments on mobile applications and through questionnaires. A daily electronic diary will be completed through the Ohmage app. The Mobility app will be used to track the patients' movement and activity. Patients will be administered a questionnaire at the 1 and 2 week endpoints.
  Interventions: Other: Electronic Diary; Other: Questionnaire

INTERVENTIONS:
Other: Electronic Diary — The electronic diary asks subjects questions about their compliance with mobile application usage. The questions contained in this diary ask patients how often their personal mobile device has been on their person, if and how long the applications relevant to the study were turned off, and why patients failed to comply with study requirements.
Other: Questionnaire — Study patients will be asked to complete a questionnaire at the 1 and 2-week endpoints. This questionnaire is administered in order to measure patient satisfaction with the mobile applications.

SUMMARY:
Mobile technology can be used to passively capture data tracing features and fluctuations of patients' daily activities, including activity levels, location patterns, sleep, and a wide variety of other health-relevant metrics. This data can then be combined with contextual recall, collected through a mobile app, to enhance passively captured behavioral data. The resulting data collection is objective, real-time, and contextual, thus addressing the pitfalls of conventional measurement of pain treatment outcomes.

DETAILED DESCRIPTION:
The goal of this pilot study is to assess the feasibility and value of using smart phone applications to collect objective, quantitative functional data from patients under active treatment for chronic pain.

35 subjects will be enrolled from the Weill Cornell Pain Medicine Center to ensure a total of 30 completed sets of surveys (15 males, 15 females). The Chronic Pain Registry (a data registry utilized to assess the outcomes of chronic pain patients) will provide data regarding the patients' demographics, diagnosis, and prescribed medications. The mobile applications ("Mobility" and "Ohmage") will be downloaded in the office with a demonstration of proper use. "Ohmage" is a data collection application, designed for use on a smart phone or tablet, and allows for both passive and active capture of data via a device's internal sensing mechanisms and through a user's participation in surveys. "Mobility" is a mobile phone sensor application, designed for both android and iPhone devices, that allows a phone to passively capture information about its user's activity. The "Mobility" application uses an activity classifier algorithm to determine if the user is stationary, walking, running, or driving based on how quickly the WiFi and/or GPS signals change, coupled with the strength of motion detected by the phone's internal accelerometer. Ohmage aggregates the Mobility application's generated data and uploads the data to a secure server for study and analysis. Patients will be asked to keep a daily electronic diary via the Ohmage app. Mobility will be used to track the patients' movement and level of activity. Telephone assistance will be available in case of technical problems (Monday to Friday, 9AM-5PM). An audible alarm reminder will be programmed to encourage compliance with use as well as timely completion of the compliance diary.

Two iterative usability cycles will be conducted with assessment of the compliance diary and questionnaire administration at the 1 and 2-week endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients with eligible smart phone devices (iPhones and Androids- working, newer models (released in the last 3 years)) running a sufficient, current version of iOS or Android
* Chronic low back pain (at least 3 months) with or without lower extremity pain (i.e. lumbar radiculopathy, spinal stenosis)
* Average pain is rated at least moderate (numerical score greater than or equal to 5/10)
* Ages 18 - 65 years
* Participating in Chronic Pain Registry (standard of care)

Exclusion Criteria:

* Conditions limiting mobility
* Non-ambulatory (wheelchair bound)
* Movement or neuromuscular disorders
* Significant lower extremity weakness
* Severe cardiorespiratory disease
* Moderate to severe cognitive impairment
* Active cancer therapy (chemotherapy or radiation) in the last year
* Major surgery in the last 3 months
* Inability to comply with study requirements per investigator judgement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study subjects will be chronic pain patients being treated for moderate to severe chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Feasibility (measured by adequate enrollment and compliance) | 2 weeks
  The primary objective is to demonstrate that this mobile technology application is feasible as . The compliance threshold for feasibility is defined as at least 50% of patients report diaries showing they had their mobile device powered on, with the app running (raw data), and the phone physically on them for a total of 12 hours per day on average. This will be calculated over the first week of data collected, second week of data, and then also the combined 2 weeks of data.

SECONDARY OUTCOMES:
Patient Satisfaction (demonstrated by questionnaires) | 2 weeks
  Measure outcomes related to the usability and patient satisfaction with the mobile application, as demonstrated by questionnaires at the 1-week and 2-week endpoints.
Compliance (reasons patients turned their phone off, or did not keep the smart phone on them) | 2 weeks
  We will explore the reasons patients turned their phone off, or did not keep the smart phone on them, all of which would be necessary for accurate data capture.
Demographics | 2 weeks
  We will analyze the population of patients who were eligible for the study but declined enrollment, as well as identifying specific subpopulations of patients who had difficulty with compliance, dropped out, or who had low satisfaction and usability scores.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Witkin, MD, Principal Investigator — Weill Cornell Medical College Department of Anesthesiology
Locations (1):
- Weill Cornell Pain Medicine Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD